CLINICAL TRIAL: NCT07392814
Title: Single-Center Phase 1 Study With Escalating Doses of Tocilizumab in Combination With Venetoclax and Azacitidine Chemotherapy in Patients With Acute Myeloid Leukemia (AML). TOCIVENA
Acronym: TOCIVENA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC25_0533; 2025-524725-41-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Leukemia Acute Myeloid - AML
Keywords: Leukemia; IL6; tocilizumab
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): * Level 1: 4 mg/kg on Day 1 of cycles 1 to 3
  * Level 2: 6 mg/kg on Day 1 of cycles 1 to 3 (starting dose for the first cohort)
  * Level 3: 8 mg/kg on Day 1 of cycles 1 to 3
  * Level 4: 4 mg/kg on Days 1 and 15 of cycles 1 to 3
  Interventions: Drug: increase dose of tocilizumab

INTERVENTIONS:
Drug: increase dose of tocilizumab — Combining tocilizumab with the standard treatment of azacitidine and venetoclax

SUMMARY:
This is a phase 1, open label, interventional, single center, in patients with Acute Myeloid Leukemia (AML). This study will investigate dose escalation of tocilizumab in combination with venetoclax and azacitidine chemotherapy.

The patient population will consist of adults men and women at least 18 years, who meet eligibility criteria. In this study we propose combining tocilizumab with the standard treatment of azacitidine and venetoclax for patients with AML who are not eligible for intensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* First-line AML regardless of karyotype and molecular profile
* ECOG <= 3
* Patient eligible for chemotherapy combining azacitidine and venetoclax
* Informed consent
* Liver function tests: transaminases < 3x normal, bilirubin < 1.5x normal
* Creatinine clearance > 30 ml/min

Exclusion Criteria:

* LAM3
* Patients eligible for intensive "3+7" treatment
* Uncontrolled infection
* Active and/or treated infection with Hep B, C, or HIV
* No social security or other health insurance
* Pregnant women or patients who cannot use contraception due to fertility
* Breastfeeding women
* Minors
* Adults under guardianship, conservatorship, or legal protection
* Hypersensitivity to any of the active substances or excipients (see SPCs)
* Patients unable to understand spoken or written French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2028-07-10 (Estimated); Study Completion 2030-07-10 (Estimated)

PRIMARY OUTCOMES:
DLT | 42 days
  number of DLT

SECONDARY OUTCOMES:
response to treatment | 28 months
  number of response
response to treatment | 28 months
  number of response without detectable residual disease
Death | 48 months
  number of days between Day 1 and Death
follow - up | 48 months
  number of days between Day 1 and follow - up date
relapse | 48 months
  number of days between remission day 1 and relapse
death | 48 months
  number of days between remission and death
follow up | 48 months
  number of days between remission and follow - up date
relapse | 48 months
  number of days between remission and relapse
relapse | 48 months
  number of relapse
neutrophil | 48 months
  number of days of neutrophil recovery
platelets | 48 months
  number of days of platelets recovery
infection | 48 months
  number of infection
cytokine | 48 months
  number of cytokine
tocilizumab | 48 months
  number of tocilizumab

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No